CLINICAL TRIAL: NCT02940535
Title: Low Dose GnRHa Early Luteal Phase Down Regulation Versus GnRHa Ultra-short Protocol for Poor Ovarian Response: a Randomized Control Trial
Brief Title: Low Dose GnRHa Early Luteal Phase Down Regulation Versus GnRHa Ultra-short Protocol for Poor Ovarian Response
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Navy General Hospital, Beijing (Other)
Responsible Party: Principal Investigator, Yunhai Chuai, Department of Obstetrics and Gynecology, Navy General Hospital, Beijing, Navy General Hospital, Beijing
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SW001
Record Dates: First submitted 2016-08-01; First posted 2016-10-21 (Estimated); Last update posted 2016-10-21 (Estimated); Status verified 2016-10

CONDITIONS: Subfertility, Female; Ovulation Disorder
MeSH Terms: conditions — Infertility, Female | interventions — Triptorelin Pamoate; Menotropins; Chorionic Gonadotropin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Low Dose GnRHa (Experimental): Diphereline 0.375mg was administered in the early-luteal-phase. Human menopausal gonadotropin/human chorionic gonadotropin (HMG/HCG) was administered start in the day 28.
  Interventions: Drug: Diphereline (Triptorelin embonate); Drug: human menopausal gonadotropin; Drug: human chorionic gonadotropin
- GnRHa Ultra-short Protocol (Active Comparator): Decapeptyl 0.1mg was administered in the menstrual day 2 to 7. Human menopausal gonadotropin/human chorionic gonadotropin (HMG/HCG) was administered start in the menstrual day 2.
  Interventions: Drug: Decapeptyl (Triptorelin); Drug: human menopausal gonadotropin; Drug: human chorionic gonadotropin

INTERVENTIONS:
Drug: Diphereline (Triptorelin embonate)
  Arms: Low Dose GnRHa
Drug: Decapeptyl (Triptorelin)
  Arms: GnRHa Ultra-short Protocol
Drug: human menopausal gonadotropin
Drug: human chorionic gonadotropin

SUMMARY:
The management of the poor responder patients is very difficult. Currently, there is no any standard treatment for poor responder patients. The study is designed to test a modified GnRHa protocol for poor ovarian response, low dose GnRHa early luteal phase down regulation, compare with GnRHa ultra-short protocol. This is a randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* At least two of the following three features must be present: i. Advanced maternal age (≥40 years) or any other risk factor for POR (poor ovarian response); ii. A previous POR (≤3 oocytes with a conventional stimulation protocol); iii. An abnormal ovarian reserve test (i.e. AFC <7 follicles or AMH <1.1 ng/ml).

Exclusion Criteria:

* Contraindications for IVF/ICSI
* Contraindications for pregnancy
* Primary ovarian insufficiency
* AFC <3
* PGD/PGS

Ages: 35 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2016-12; Primary Completion 2019-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
live birth | 3 years
  The event that a FETUS is born alive with heartbeats or RESPIRATION regardless of GESTATIONAL AGE. Such liveborn is called a newborn infant (INFANT, NEWBORN).

SECONDARY OUTCOMES:
clinical pregnancy rate | 3 years
  Presence of fetal heart at transvaginal ultrasound at 6 weeks of gestation or 6 weeks after starting the intervention.

OTHER OUTCOMES:
multiple pregnancy | 3 years
  The condition of carrying two or more FETUSES.
miscarriage | 3 years
  Expulsion of the product of FERTILIZATION before completing the term of GESTATION and without deliberate interference.
Ectopic pregnancy | 3 years
  A potentially life-threatening condition in which EMBRYO IMPLANTATION occurs outside the cavity of the UTERUS. Most ectopic pregnancies (>96%) occur in the FALLOPIAN TUBES, known as TUBAL PREGNANCY. They can be in other locations, such as UTERINE CERVIX; OVARY; and abdominal cavity (PREGNANCY, ABDOMINAL).
Dose of HMG required | 3 years
Duration of HMG stimulation | 3 years
Number of oocytes retrieved | 3 years
Number of embryos obtained | 3 years
Number of embryos frozen | 3 years
Adverse effects | 3 years
  According to the Common Terminology Criteria for Adverse Events, version 4.0 (CTCAE 2009). Some adverse events will be studied as separate outcomes, including ovarian hyperstimulation syndrome (OHSS).
Congenital Abnormalities | 3 years
  Malformations of organs or body parts during development in utero.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Shang, Dr, Principal Investigator — Navy General Hospital, Beijing; Yunhai Chuai, Dr, Principal Investigator — Navy General Hospital, Beijing; Mingming Shu, Dr, Principal Investigator — Navy General Hospital, Beijing; Ming Zhou, Dr, Principal Investigator — Navy General Hospital, Beijing; Huiming Han, Dr, Principal Investigator — Navy General Hospital, Beijing; Mengnan Chen, Dr, Principal Investigator — Navy General Hospital, Beijing; Lei Chen, Principal Investigator — Navy General Hospital, Beijing
Locations (1):
- Navy General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Siristatidis CS, Yong LN, Maheshwari A, Ray Chaudhuri Bhatta S. Gonadotropin-releasing hormone agonist protocols for pituitary suppression in assisted reproduction. Cochrane Database Syst Rev. 2025 Jan 9;1(1):CD006919. doi: 10.1002/14651858.CD006919.pub5. PMID 39783453